CLINICAL TRIAL: NCT00763984
Title: PERL 4: Promoting Effective Recovery From Labor
Brief Title: Self-Care to Prevent Birth-Related Urinary Incontinence in Diverse Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Carolyn Sampselle, Carolyne K. Davis Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2R01NR007618-06A1 (NIH); 2R01NR007618 (NIH); 2R01NR007618-06A1 (NIH); HUM00015712 (Other: University of Michigan IRB); NCT00763984 (Registry Identifier: ClinicalTrials.govID)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Urinary Incontinence
Keywords: Bladder Control for Women; Exercising Your Pelvic Muscles; Kegel Exercises: How to Strengthen Pelvic Floor Muscles; Kegel Exercises for Your Pelvic Muscles; Pelvic Floor Disorders; Pelvic Support Problems; Pregnancy; Pregnancy Childbirth and Bladder Control; Urinary Incontinence; Urinary Incontinence: Embarrassing but Treatable
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Usual Care (Active Comparator): This group will receive routine care, however, it is possible that that control condition participants will receive Pelvic Floor Muscle Training (PFMT) instruction from their health care providers. We will monitor control women's knowledge, adoption and maintaining of PFMT
  Interventions: Behavioral: Usual Care
- 2 Bladder Health Class (Experimental): Modeled on our intervention with older women, Bladder Health Class (BH Class) will include Pelvic floor muscle training (PFMT), defined by the International Continence Society as repetitive selective voluntary contraction and relaxation of specific pelvic floor muscles, and bladder training (BT), defined as a program of scheduled voiding with gradually progressive voiding intervals. The BT instructions will be modified for this pregnant group. We will monitor control women's knowledge, adoption and maintaining of PFMT and BT.
  Interventions: Behavioral: Bladder Health class

INTERVENTIONS:
Behavioral: Usual Care — This group will receive routine care, however, it is possible that that control condition participants will receive Pelvic Floor Muscle Training (PFMT) instruction from their health care providers. We will monitor control women's knowledge, adoption and maintaining of PFMT.
  Arms: 1 Usual Care
Behavioral: Bladder Health class — Modeled on our intervention with older women, Bladder Health Class (BH Class) will include Pelvic floor muscle training (PFMT), defined by the International Continence Society as repetitive selective voluntary contraction and relaxation of specific pelvic floor muscles, and bladder training (BT), defined as a program of scheduled voiding with gradually progressive voiding intervals. The BT instructions will be modified for this pregnant group. We will monitor control women's knowledge, adoption and maintaining of PFMT and BT.
  Arms: 2 Bladder Health Class

SUMMARY:
The primary goal of this project is to determine the efficacy of an antenatal Bladder Health class to prevent UI in a diverse sample of African American, Caucasian, and Hispanic childbearing women. The determination of efficacy will be made at 12-months post index birth, a time point that is a traditional benchmark of recovery from childbirth, using UI incidence/severity as the primary outcome.

DETAILED DESCRIPTION:
This study is significant because UI prevalence is 34% overall among US women, nearly half of whom consider their incontinence to be moderately to extremely bothersome. UI is 2.0 to 2.6 fold greater in women after pregnancy and childbirth as compared to their never pregnant counterparts, with the incidence increasing after each child. UI impact increases as women age extending into middle and later life. The financial cost of UI in the United States exceeds $19 billion per year . Other costs are identified in the Healthy People 2010 report 22 and include: 1) decreased activity/ fitness, which can be seriously affected because women who are concerned about accidental leakage markedly curtail physical activity and 2) increased depression, which has been linked to UI in women. Women are at least twice as likely as men to have UI; pregnancy and childbirth are major explanatory factors. In perimenopausal women, prevalence of any UI was 57% and of moderate to severe UI was 25%; after controlling for age, race/ethnicity, menopausal status and body mass index, parity persisted as a significant predictor of UI with an OR of 1.62 (CI 1.31, 2.01).

Noninvasive interventions during the period of childbearing are of particular interest for UI prevention in women. Two self-management practices recommended for the initial treatment of UI are: Pelvic floor muscle training (PFMT), defined by the International Continence Society as repetitive selective voluntary contraction and relaxation of specific pelvic floor muscles, and bladder training (BT), defined as a program of scheduled voiding with gradually progressive voiding intervals. The Knack Maneuver (a preemptive pelvic floor muscle contraction to decrease stress UI and/or suppress urge UI) has demonstrated efficacy in older women diagnosed with UI. In childbearing women, only PFMT has been tested with a rigorous RCT design. We taught PFMT, the Knack, and BT as a combined strategy to older women and found a two-fold prevention effect. The proposed project is innovative because it will be the first to our knowledge to test the preventive capacity of an intervention in childbearing women that combines PFMT, the Knack, and BT. This project is also innovative because it will be conducted with a diverse sample of primiparous/multiparous women, using a 3-year follow-up period. Because PFMT is the only self-management strategy that is currently recommended practice for maternity patients, we will use PFMT adherence in comparisons between the treatment and control conditions

Recruitment and Informed Consent:

Fliers specifying eligibility criteria and benefits of research participation will be prominently displayed in the waiting areas and in the women's bathrooms of the respective clinical sites. Potential participants will be invited to speak with a designated site-based contact re: what participation in the study would entail. This individual will answer initial questions, review written material that describes study participation, conduct verbal screening, and obtain informed consent from eligible individuals. Eligible participants will be scheduled for a clinic visit at the respective site for a clinic visit to obtain clinical verification of no objective incontinence (negative standing stress test) and evidence of ability to contract the pelvic floor correctly (digital measure). Following determination of eligibility, participants will be randomized into control (routine care) or treatment (scheduled for Bladder Health class) condition.

ELIGIBILITY:
Inclusion Criteria:

Women who are pregnant and expecting their first, second, or third baby are eligible if they:

* are age eighteen years or older
* are able to understand and read English or Spanish
* are low risk antepartum (first, second or third pregnancy)
* are 16-25 weeks pregnant
* expect a vaginal birth
* have lost no more than a few drops of urine as often as every other day
* have no previous or current urinary incontinence treatment with medication, formal behavioral programs or surgery
* have no history of bladder cancer, diabetes, stroke, multiple sclerosis, muscular dystrophy, cerebral palsy, Parkinson's, epilepsy, or trauma of the spinal cord
* Do not have (or have not had within the last 3 years) *chronic urinary tract infection. *Chronic is defined as having more than 3 urinary tract infections in one year.

Exclusion Criteria:

* If participant does not meet all of the above criterion for inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
UI incidence/severity | 12 months - 3 years post-index birth

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Sampselle, PhD RNC FAAN, Principal Investigator — University of Michigan, School of Nursing, Grants and Research Office
Locations (3):
- United States (3):
  - University of Michigan Health System, Ann Arbor, Michigan
  - Jackson Center for Family Health, Jackson, Michigan
  - La Clinica de la Santa Teresa, Pontiac, Michigan

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735